CLINICAL TRIAL: NCT01320059
Title: A Phase I Study of 18F-Fluoro-PEG6-IPQA as a PET Imaging Agent for Active/Mutant EGFR Expression in Tumors
Brief Title: Study of 18F-Fluoro-PEG6-IPQA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-0832; W81XWH-05-2-0027 (Other: DOD); NCI-2014-01375 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: 18F-Fluoro-PEG6-IPQA; Radioactive Imaging Solution; Non-Small Cell Lung Cancer; Positron Emission Tomography; PET Scan; CT; Computed Tomography
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — 4-((3-iodophenyl)amino)-7-(2-(2-(2-(2-(2-(2-(18F)fluoroethoxy)ethoxy)ethoxy)ethoxy)ethoxy)ethoxy)quinazoline-6-yl-acrylamide; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging with 18F-PEG6-IPQA (Experimental): Radioactive injection given by vein before multiple (3) PET scans.
  Interventions: Drug: 18F-PEG6-IPQA; Procedure: Positron emission tomography (PET)

INTERVENTIONS:
Drug: 18F-PEG6-IPQA — Radioactive injection (PET imaging agent) given by vein before PET scans.
Procedure: Positron emission tomography (PET) — 3 PET scans performed after injection and positioning CT. Imaging should take about 3 hours.
  Other Names: PET; Imaging

SUMMARY:
The goal of this clinical research study is to learn if an imaging solution called 18F-PEG6-IPQA can help to find tumors when used in positron emission tomography (PET) scans. The safety of the solution and how the solution is processed by your body will also be studied.

DETAILED DESCRIPTION:
18F-PEG6-IPQA is a solution that is designed to be attracted to tumor cells. The imaging solution has a small dose of radiation added to it, which may help doctors see the cancer cells better during imaging scans. This is the first study using 18F-PEG6-IPQA in humans.

Study Imaging:

If you are found to be eligible to take part in this study, you will visit the clinic on Day 1 for the injection of the study solution and PET scans. This imaging study will be performed at FDA-cleared PET-CT scanners at MD Anderson sites, including at the Center for Advanced Biomedical Imaging (CABI).

For up to 6 hours before the PET scans and computed tomography (CT) scans, you must not eat or drink anything except water. This is called fasting.

A small tube will be placed in your arm and you will receive an injection of 18F-PEG6-IPQA.

After the injection, scanning will begin immediately. You will have 3 PET scanning sessions with a PET/CT scanner. Before each PET scan, you will have a CT scan to make sure you are in the right position for the PET scans. Each PET scan may last up to 1 hour. Each positioning CT scan should take about 5 minutes. You will have a 10 minute "rest period" between each PET scan.

Study Visits:

On Day 1:

* Before the imaging solution is injected, your vital signs and an ECG rhythm strip will be collected. The study staff will insert an intravenous (IV) needle and line into each of your arms.
* Right after the injection of the study drug, blood (about 2 tablespoons total) will be drawn for pharmacokinetic (PK) testing from one of the existing IV lines. PK testing measures the amount of study solution in the body at different time points. Blood will be drawn at 1, 3, 8, 16, 30, 45, 60, 90, and 150 minutes after the injection of 18F-PEG6-IPQA for a total of 9 draws.
* About 30 minutes after the injection, your vital signs will be measured and the injection site will be checked.
* Urine will be collected during the 10 minute rest periods in between scans or at the completion of the 3-hour scanning period.
* After the scans are completed (about 3 hours after the injection) your vital signs and injections site will be checked again, and you will have an ECG rhythm strip taken. Blood (about 2 tablespoons) and urine will also be collected for routine tests.

On Days 2 and 7:

* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* Your vital signs and the injection site will be checked
* You will be asked about any side effects you may be having since the injection.

End-of-Study Visit:

The end-of-study visit will be about 14 days after the injection of 18F-PEG6-IPQA and imaging scans. The following tests and procedures will be performed:

* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* You will have a physical exam, including measurement of your vital signs.
* The injection site will be checked.
* You will have an ECG.

Length of Study:

You will be in this study for about 14 days. You will be taken off study early if intolerable side effects occur.

This is an investigational study. 18F-PEG6-IPQA is not FDA-approved or commercially available for use in imaging scans. Its use in this study is investigational.

The scans performed with 18F-PEG6-IPQA are also considered investigational and will not be used for planning any of your future cancer treatment.

Up to 15 patients will take part in this study. All participants will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must give written informed consent
2. Patients should have pathologically or cytologically confirmed Stage IV non-small cell lung cancer with clinical or radiological evidence that it is not amenable to therapy with curative intent. Prior EGFR tyrosine kinase inhibition (TKI) therapy is permitted but not required.
3. Patients should be potential candidates for therapy with an EGFR tyrosine kinase inhibitor or with an anti-EGFR monoclonal antibody by clinical criteria.
4. Patients should have clinical characteristics that would suggest an increased probability of benefit from an EGFR inhibitor. Specifically, they should have known EGFR mutations or high gene copy number.
5. Patients should have at least one tumor deposit that is > 1.0 cm in diameter, and that is amenable to imaging
6. Patients should be Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Patients with brain metastases are eligible provided they meet all other eligibility criteria and do not require corticosteroids or enzyme-inducing anticonvulsants and provided it is felt clinically that they will not require radiotherapy in the three (3) weeks subsequent to their participation in the study
8. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately. The patient, if a man, agrees to use effective contraception or abstinence
9. The patient must be considered legally capable of providing his or her own consent for participation in this study
10. Subjects must be at least 18 years of age

Exclusion Criteria:

1. Radiotherapy, chemotherapy or any investigational agent within the previous 2 weeks of administrating 18F-PEG6-IPQA for PET/CT imaging.
2. A non-investigational targeted agent within the previous 2 weeks of 18F-PEG6-IPQA for PET/CT imaging.
3. Thoracic or abdominal surgery within the previous 2 weeks of 18F-PEG6-IPQA for PET/CT imaging.
4. A tumor that is known to have a K-ras mutation
5. Squamous cell, large cell undifferentiated, neuroendocrine or small cell undifferentiated carcinoma of the lung
6. A known other currently active malignancy. (Benign tumors and benign polyps, basal cell carcinomas of skin, superficial papillary bladder tumors, and pre-invasive carcinoma of the cervix are permitted)
7. Physical inability to undergo a scanning procedure (e.g., inability to lie flat for the required period of time - three sessions of roughly an hour each with ten minutes' rest in between)
8. Serum creatinine >1.5 x upper limit of normal (ULN), bilirubin >1.5 x ULN, AST > 3 x ULN
9. 10. Hemoglobin < 8 g/dL, absolute neutrophil count < 1,500/mm3, platelet count <100,000/mm3
10. Potentially life-threatening arrhythmia; myocardial infarct within the previous 3 months; unstable angina, or angina at rest; congestive heart failure (New York Heart Association Functional Classification class II or worse), uncontrolled hypertension (systolic BP > 160 or diastolic BP >100).
11. Active acute infection (i.e. currently treated with antibiotics). Patients with chronic infections such as hepatitis B or C, mycobacterium avium or similar infections will be eligible provided they meet all other eligibility criteria.
12. Oxygen saturation <90% on room air
13. Clinical requirement for systemic corticosteroids for control of cerebral edema or for enzyme-inducing anticonvulsants. (Inhaled steroids and systemic steroids for chronic obstructive pulmonary disease (COPD) are permitted).
14. Pregnant or nursing
15. Any condition that is unstable or could jeopardize the safety of the patient and his or her compliance in the study, in the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Optimum dosimetry of 18F-PEG6-IPQA sodium injection based on critical organ safety | Safety measurements performed from administration of injection until 2 weeks after administration.
  Optimum dosimetry of 18F-PEG6-IPQA injection for each cohort derived from previous cohort based on statistical evaluation of critical organ exposure and safety limitations. Safety measurements performed from administration of 18F-PEG6-IPQA injection until 2 weeks after administration. The biodistribution of 18F-PEG6-IPQA will be measured during positron emission tomography (PET) scans. The percent injected dose (%ID) obtained in different organs will be derived from the PET data.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Podoloff, MD,BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org